CLINICAL TRIAL: NCT01253356
Title: A Multicenter, Randomized, Controlled Pilot Study of Intra-Aortic Balloon Counterpulsation to Prevent Perioperative Cardiac Events in High-Risk Cardiac Patients Undergoing Noncardiac Surgery
Brief Title: ACTIONS - Aortic Counterpulsation to Improve Outcomes in Noncardiac Surgery
Acronym: ACTIONS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Only 1 patient recruited and deemed ineligible.
Sponsor: Datascope Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P-00002
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Patients With History of Ischemic Heart Disease With LV Dysfunction Undergoing Noncardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No IABP (No Intervention): Standard of care and no IABP
- Intra-Aortic Balloon Pump (IABP) (Active Comparator): Standard of care, IABP inserted < or = 3 hours before noncardiac surgery, maintained for > or = 12-24 hours after surgery
  Interventions: Device: IABP

INTERVENTIONS:
Device: IABP — Insertion of intra-aortic balloon < or = 3 hours before noncardiac surgery and maintained > or = 12-24 hours after surgery
  Arms: Intra-Aortic Balloon Pump (IABP)

SUMMARY:
The use of the IABP, in addition to standard care, in high-risk cardiac patients undergoing major noncardiac surgery is feasible and may result in improved perioperative outcomes at 30 days compared with standard care alone, while maintaining acceptable safety with respect to vascular accesss-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years with planned elective major abdominal, noncardiac thoracic, head and neck, vascular, or orthopedic surgery and guideline-treated iscehmic heart disease with left ventricular dysfunction (systolic ejection fraction < or = 30%)

Exclusion Criteria:

* Unstable coronary syndromes Decompensated or NYHA Class IV heart failure Hemodynamic instability Cardiac biomarker instability Need for surgical procedure interfering with placement of IABP Cardiogenic shock Septic shock Contraindication to IABP use Clinical need for IABP ASA score > or = 5 Pregnancy Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Safety | 30 days
  Amputation, Clinically significant bleeding, Vascular complications

SECONDARY OUTCOMES:
Efficacy | 30 days
  A composite of the following:
  All-cause mortality, Cardiovascular mortality, Hemorrhagic or ischemic stroke, New nonfatal myocardial infarction, New or worsening congestive heart failure, Hemodynamically significant arrhythmia requiring intervention

CONTACTS AND LOCATIONS:
Overall Officials: Don Poldermans, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Genesis Medical Center, Davenport, Iowa, United States